CLINICAL TRIAL: NCT03112343
Title: An Information and Communication Technology-based Centralized Clinical Trial to Determine the Efficacy and Safety of Insulin Dose Adjustment Education Based on a Smartphone Personal Health Record Application
Brief Title: Information and Communication Technology Based Centralized Clinical Trial Monitoring System for Insulin Dose Adjustment
Acronym: ICT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Ministry of Trade, Industry & Energy, Republic of Korea (Other Government); Korea Evaluation Institute of Industrial Technology (Other); Daegu Metropolitan City, Korea (Other Government); ICT Clinical Trial Coordination Center (Other)
Responsible Party: Principal Investigator, Sang-Man Jin, Assistant professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-08-006-001
Record Dates: First submitted 2017-04-04; First posted 2017-04-13 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus; Insulin Hypoglycemia; Insulin-dependent Diabetes Mellitus
Keywords: ICT based clinical trial; Contract research organization (CRO); eCRF; Joint Electronic-institutional review board (eIRB); Centralized monitoring
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Health Records, Personal

STUDY DESIGN:
Intervention Model Description: randomized in a 1:1 ratio to either the information and communication technology(ICT)-based intervention group or the conventional intervention group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICT-based intervention (Active Comparator): Subjects in the ICT-based intervention group have algorithm-based feedback messages in addition to conventional intervention
  Interventions: Device: Algorithm-based feedback messages; Device: Personal Health Record
- Conventional intervention group (Placebo Comparator): Subjects in the conventional intervention group will only save and send their health information to the server via the personal health record app
  Interventions: Device: Personal Health Record

INTERVENTIONS:
Device: Algorithm-based feedback messages — ICT-based intervention group have algorithm-based feedback messages in addition to conventional intervention
  Arms: ICT-based intervention
Device: Personal Health Record — Subjects will save and send their health information to the server via the personal health record app

SUMMARY:
This is a 24-week, open-label, randomized, multi-center trial conducted in three tertiary hospitals. There are three follow-up measures; at baseline, post-intervention at Week 12, and Week 24. Subjects are diagnosed as type 1 DM, type 2 DM, and/or post-transplant DM, and initiate or currently use insulin therapy. After the given education on insulin dose titration and prevention for hypoglycemia and 1 week of run-in period, subjects are randomized in a 1:1 ratio to either the ICT-based intervention group or the conventional intervention group. Subjects in conventional intervention group will save and send their health information to the server via the PHR app, whereas those in ICT-based intervention group have additional algorithm-based feedback messages. The health information includes levels of blood glucose, insulin dose, details on hypoglycemia, food diary, and number of steps. The primary outcome will be the proportion of patients who reach an optimal insulin dose within 12 weeks of enrolling in the study without severe hypoglycemia or unscheduled clinic visits.

This study is based upon work supported by the Ministry of Trade, Industry & Energy (MOTIE, Korea) under Industrial Technology Innovation Program (No. 10059066, 'Establishment of ICT Clinical Trial System and Foundation for Industrialization.")

DETAILED DESCRIPTION:
This is a 24-week, open, randomized, multi-center ICT-based clinical trial conducted in three different hospitals including Samsung Medical Center, Kangbuk Samsung Hospital, and Samsung Changwon Hospital. There are three follow-up measures; at baseline, post-intervention at Week 12, and Week 24. Subjects diagnosed as T1DM, T2DM, and/or post-transplant DM who initiate or currently use insulin therapy will be given education on insulin injection, dose adjustment, and prevention for hypoglycemia and provided at-home measurement device at Visit 1 for screening. Subjects will receive instructions to check daily glucose levels by home glucose meter, to record insulin regimen and dose, the hypoglycemia diary if blood glucose <70 mg/dL or a hypoglycemic event occurs in the apps, and to synchronize data for automatically transferring to system. Subjects who synchronized their information more than once during 1 week of run-in period will be selected into clinical trial and randomly assigned to either ICT-based intervention group or conventional intervention group at a ratio of 1:1. After the randomization, at Week 1, diabetes educators provide telephone counselling for re-instructing insulin dose adjustment and for re-confirming their use of at-home measurement device and PHR apps at Visit 2 (televisit). Subjects in ICT-based intervention group will have algorithm-based feedback messages when their glucose levels are out of ranges, in addition to recording, saving and sending their data to the server via the PHR app, and those in conventional intervention group will only record, save and send their data to the server via the PHR app. Investigators examine the saved health information such as levels of blood glucose, insulin dose, details on hypoglycemia recorded in hypoglycemia diary, food diary, and number of steps transferred through PHR apps. At each clinical visit, anthropometric parameters, current medication use including types of insulin, insulin dose, and other glucose-lowering agents, vital signs, body composition, and questionnaire for satisfaction investigation are examined face-to-face, and blood tests are performed. The unscheduled visit to clinic could be applied if a subject has one or more severe hypoglycemia (requiring other help for recovery) during the study period, or hypoglycemia (<70 mg/dL) twice or more times per week, or fasting blood glucose >200 mg/dL three or more times in the morning, and wants to see a doctor during Week 1-12. The unscheduled visit to clinic is also allowed to the subjects who have difficulty in insulin dose adjustment despite of two or more unscheduled tele-visit. However, even if this criterion does not apply, patients who initiate insulin or change their regimen (eg, from basal insulin once daily to premixed insulin or multiple dose insulin injections) will be allowed to have additional planned doctor visits prior to Visit 3, which is not included in the unscheduled visit, but will be evaluated as scheduled additional visit. The primary outcome will be the proportion of patients who reach an optimal insulin dose within 12 weeks of enrolling in the study without severe hypoglycemia or unscheduled clinic visits.

ELIGIBILITY:
Inclusion Criteria

1. age between 18-69 years
2. diagnosis of T1DM, T2DM, and/or post-transplant DM (Post-transplant DM includes both diagnosed T1DM or T2DM before organ transplantation and first diagnosed DM after organ transplantation)
3. initiation or current use of insulin therapy including once-daily basal insulin (including basal insulin only or basal insulin plus rapid-acting insulin), premixed insulin, or NPH)
4. most recent hemoglobin A1c (HbA1c) ≥7.0% based on the National Glycohemoglobin Standardization Program (NGSP) at least 3 months prior to participation (recent HbA1c values measured <3 months prior to screening are permitted.)
5. available to use smartphone and wireless internet
6. Voluntarily write consent to participate in the trial

Exclusion criteria

1. on insulin pump
2. history of alcohol or drug abuse 1 year prior to participation
3. history of psychological disorder (e.g., schizophrenia, depression, or bipolar disorder)
4. history of severe visual or hearing impairment
5. pregnant
6. any condition, in the investigator's opinion, not suitable for enrollment eligibility.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
the proportion of patients who reach his/her optimal insulin dose within 12 weeks of enrolling in the study without severe hypoglycemia or unscheduled clinic visits. | Week 12
  Reaching optimal insulin dose: A.For a patient who uses basal insulin only or basal insulin with pre-meal rapid-acting insulin once per day,1)3 or more fasting blood glucose(FBG) values in the morning within the target range(80-130mg/dL or 100-140 mg/dL) during Week12,2)no nocturnal(11pm-7am) or pre-breakfast hypoglycemia(<70mg/dL) during Week12,3)variation of basal insulin dose (the difference between the highest and lowest basal insulin dose) of <10% of mean total basal insulin dose during Week12. B.For a patient who uses MDI at least twice per day, the criteria A plus 4)3 or more days in which correction dose premeal insulin is required less than 3times per day during the Week12,5) no daytime(7am-11pm) hypoglycemia during Week12. C.For a patient who uses premixed insulin or NPH,1)3 or more FBG values in the morning and evening within the target range during Week 12,2) no nocturnal or pre-breakfast hypoglycemia during Week12

SECONDARY OUTCOMES:
the proportion of patients who reach HbA1c <7% without severe hypoglycemia (unrecoverable hypoglycemia without the help of others) at Week 24 | Week 24
  the proportion of patients who reach HbA1c <7% without severe hypoglycemia (unrecoverable hypoglycemia without the help of others) at Week 24
the proportion of patients who reach HbA1c <7% without severe hypoglycemia (unrecoverable hypoglycemia without the help of others) at Week 12 | Week 12
  the proportion of patients who reach HbA1c <7% without severe hypoglycemia (unrecoverable hypoglycemia without the help of others) at Week 12
mean fasting blood glucose values for three consecutive days prior to Week 12 and Week 24 | Week 12 and 24
  mean fasting blood glucose values for three consecutive days prior to Week 12 and Week 24
levels of HbA1c at Week 12 and Week 24 | Week 12 and Week 24
  levels of HbA1c at Week 12 and Week 24
lipid profile at Week 12 and Week 24 | Week 12 and 24
  lipid profile at Week 12 and Week 24
the proportion of patients having hypoglycemia (total, asymptomatic, daytime, nighttime, severe hypoglycemia, and coma/convulsions) at Week 12 and Week 24 | Week 12 and Week 24
  the proportion of patients having hypoglycemia (total, asymptomatic, daytime, nighttime, severe hypoglycemia, and coma/convulsions) at Week 12 and Week 24
the number of steps during Week 1-12 and Week 13-24 | Week 12 and Week 24
  the number of steps during Week 1-12 and Week 13-24
recorded exchange unit by food group | Week 12 and 24
  recorded exchange unit by food group (grains, meats and protein, fruits, vegetables, dairy, and fats and oils) in each breakfast, lunch, and dinner on 3-day food diary at Week 12 and 24
daily insulin dose | Week 12 and Week 24
  daily insulin dose at Week 12 and Week 24
blood pressure | Week 12 and Week 24
  blood pressure at Week 12 and Week 24
body weight | Week 12 and Week 24
  body weight at Week 12 and Week 24
lean body mass | Week 12 and 24
  lean body mass at Week 12 and Week 24
fat mass | Week 12 and 24
  fat mass at Week 12 and Week 24
Satisfaction evaluation by questionnaire for ICT-based centralized clinical trial monitoring | Week 12 and 24
  Satisfaction evaluation by questionnaire for ICT-based centralized clinical trial monitoring at Week 12 and 24
Satisfaction evaluation by DTSQ | Week 12 and 24
  Satisfaction evaluation by DTSQ at Week 12 and 24
the number of telephone counselling by diabetes educators | Week 12 and 24
  the number of telephone counselling by diabetes educators
the number of self-monitoring blood glucose measurements | Week 12 and 24
  the number of self-monitoring blood glucose measurements

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Man Jin, MD PhD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim G, Bae JC, Yi BK, Hur KY, Chang DK, Lee MK, Kim JH, Jin SM. An information and communication technology-based centralized clinical trial to determine the efficacy and safety of insulin dose adjustment education based on a smartphone personal health record application: a randomized controlled trial. BMC Med Inform Decis Mak. 2017 Jul 18;17(1):109. doi: 10.1186/s12911-017-0507-4. PMID 28720103